CLINICAL TRIAL: NCT04195152
Title: Investigation of the Incidence of Lingual Nerve Injury and Related Factors in Patients With Difficult Intubation
Brief Title: Lingual Nerve Injury in Patients With Difficult Intubation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Zeynep Nur Orhon, Principal Investigator, Istanbul Medeniyet University
Other Study IDs: İstanbulMUzeynep
Record Dates: First submitted 2019-12-04; First posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Difficult Intubation; Lingual Nerve Injuries
Keywords: Difficult intubation; Lingual nerve injury; Body mass index
MeSH Terms: conditions — Lingual Nerve Injuries | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Difficult intubation group: An intubation is called difficult if a normally trained anesthesiologist needs more than 3 attempts or more than 10 min for a successful endotracheal intubation.
  Interventions: Other: Observational
- Non difficult intubation group: An intubation is called non difficult if a normally trained anesthesiologist needs only one attempt for a successful endotracheal intubation.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — No intervention

SUMMARY:
The aim of this study is to investigate the incidence of lingual nerve injury and related factors in difficult intubation cases.

Demographic data of difficult intubation cases and body mass indices, thyromental and sternomental distances, mallampati classification, neck circumference, maximum mouth opening be recorded.Numbness of the tongue and metallic taste will be questioned

DETAILED DESCRIPTION:
The lingual nerve is the anterior descending branch of the posterior trunk of the mandibular division of the trigeminal nerve.

Lingual nerve injury is a recognised complication of orotracheal intubation and has been associated with forceful laryngoscopy.

Although left-sided neuropraxia has been reported, right-sided lesions are thought to be more common because the standard Macintosh laryngoscope exerts pressure on the right side of the tongue.

Lingual nerve injury following orotracheal intubation was first described in 1971 by Teichner who reported a right-sided neuropraxia which was attributed to direct pressure from the laryngoscope.

ELIGIBILITY:
Inclusion Criteria:

All adult patients undergo general anesthesia who have difficulty in intubation will be included in the study. The same number of patients without intubation difficulties will be included in the study as a control group.

Exclusion Criteria:

1. Patients who are not intubated under general anesthesia
2. Patients undergoing regional anesthesia or peripheral nerve block
3. Patients with laryngeal mask placed will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients undergo general anesthesia who have difficulty in intubation will be included in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of lingual nerve injury | 1 year
  The frequency of lingual nerve injury in patients with difficult intubation seen in one year period will be determined.

SECONDARY OUTCOMES:
Rate of emergency tracheotomy | 1 year
Incidence of cardiovascular complications | 1 year
Percentage of patients with teeth injuries | 1 year
Percentage of patients with oral mucosa injuries | 1 year
Percentage of patients with temporary difficulty in swallowing | 1 year
Percentage of patients with temporary difficulty in breathing | 1 year
Incidence of inability to taste | 1 year
Incidence of numbness in the tongue | 1 year
Percentage of patients with metallic taste in the tongue | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul MU Goztepe Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided